CLINICAL TRIAL: NCT01818726
Title: Open-label Study of Exjade in the Treatment of Transfusion-dependent Iron Overload in Aplastic Anemia Patients Undergoing Treatment Programs in Comparison With Control Group
Brief Title: Safety and Efficacy of Exjade in the Treatment of Transfusion-dependent Iron Overload in Aplastic Anemia Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Failure to meet the schedule of patient recruitment
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CICL670ARU02
Record Dates: First submitted 2013-03-05; First posted 2013-03-26 (Estimated); Results first posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-07

CONDITIONS: Aplastic Anemia
Keywords: Aplastic anemia; deferasirox; ICL670; renal function; transfusion-dependent iron overload; immunosuppressive treatment; Cyclosporine A; unosuppressive treatment without chelation therapy
MeSH Terms: conditions — Anemia, Aplastic | interventions — Deferasirox; Chelating Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serum ferritin level ≥ 1,000 μg/l (Experimental): Transfusion-dependent adult patients with AA and serum ferritin ≥ 1000 mg/L on programmed immune suppressive treatment with cyclosporine A who were receiving chelation with Exjade (deferasirox) during the study
  Interventions: Drug: ICL670; Drug: Chelation
- Serum ferritin level < 1,000 μg/l (Experimental): Transfusion-dependent adult patients with AA and serum ferritin < 1,000 mg/L on programmed immune suppressive treatment with cyclosporine A who were not receiving the investigational product
  Interventions: Drug: No chelation

INTERVENTIONS:
Drug: ICL670 — ICL670 was supplied in registered packages as 250mg or 500mg dispersible tablets.
  Other Names: Deferasirox
  Arms: Serum ferritin level ≥ 1,000 μg/l
Drug: Chelation — Main group of patients with aplastic anemia and transfusion-dependent iron overload underwent treatment programs of standard immunosuppressive treatment (immunosupressant - Cyclosporine A) and received chelation with ICL670 (deferasirox).
  Arms: Serum ferritin level ≥ 1,000 μg/l
Drug: No chelation — Comparative group of patients with aplastic anemia and transfusion-dependent iron overload underwent treatment programs of standard immunosuppressive treatment ( immunosupressant -Cyclosporine A)
  Arms: Serum ferritin level < 1,000 μg/l

SUMMARY:
Evaluated Exjade efficacy and safety in patients with aplastic anemia and transfusion-dependent iron overload, undergoing treatment programs of immunosuppressive treatment (Cyclosporine A) , in comparison with a group of patients undergoing treatment programs of immunosuppressive treatment (Cyclosporine A) without chelation therapy.

DETAILED DESCRIPTION:
The secondary endpoints that were originally planned for this study were not analyzed as the study ended prematurely.

ELIGIBILITY:
Inclusion Criteria:

* Main diagnosis: aplastic anemia
* Absence of severe and/or uncontrolled comorbidities
* Confirmed iron overload (serum ferritin ≥ 1000 mkg/L)
* Serum creatinine is not higher than the upper limit of normal for the given age
* Absence of severe proteinuria. Protein/Creatinine ratio should be < 0.5 mg/mg
* Liver enzymes are < 5 ULN
* Completion of a scheduled cycle of immunosuppressive treatment program, with no severe infectious or generalized hemorrhagic complications
* WHO (ECOG) performance status ≤ 2

Exclusion Criteria:

* No signed informed consent form
* Patient is under 18 years old
* Severe concomitant condition
* Severe infectious and generalized haemorrhagic complication following regular planned cycle of programmed immune suppressive treatment.
* History of increased sensitivity to active substance and any other ingredient of the medicinal product.
* Creatinine clearance (CC) < 60 ml/min and/or creatinine concentration in blood serum is 2 or more times higher than upper limit of age normal by results of 2 tests at Visits 1 and 2.
* Severe liver disorders (class C by Child-Pugh scale).
* Patients with aplastic anaemia in which chelator treatment will be ineffective due to rapid progression of the disease.
* Significant proteinuria basing on protein creatinine ratio > 1.0 mg/ml in urine sample from second urination at Visits 1 and 2 (or as an alternative in 2 of 3 urine samples at screening);
* Rare hereditary disorders related to galactose intolerance, severe deficit of lactase or glucose-galactose malabsorption;
* Pregnancy, lactation;
* Level of liver enzymes higher than 5 upper limits of age normal at Visits 1 and 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2016-10-17 (Actual); Study Completion 2016-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Estimated number of patients was 25; the actual number of patients enrolled in the study and included in efficacy analysis was 15.
Pre-assignment Details: The study enrolled adult transfusion-dependent patients with Aplastic Anaemia (AA) on programmed immune suppressive treatment.
Period: Overall Study
Arm/Group | Serum Ferritin Level ≥ 1,000 μg/l | Serum Ferritin Level < 1,000 μg/l
Started | 10 | 5
Completed | 4 | 3
Not Completed | 6 | 2
Not completed — Administrative reasons | 5 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Decision to perform 2nd course of trtmnt | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all enrolled patients received at least one dose of the investigational product, as well as all patients from the comparison group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Serum Ferritin Level ≥ 1,000 μg/l | Serum Ferritin Level < 1,000 μg/l | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.0 (9.33) | 37.0 (10.10) | 35.0 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 1 | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Ferritin Values
Description: Change from baseline was be summarized descriptively for all on-treatment study visits.
  Changes to the planned statistical analysis were related to significant withdrawal of patients from the Per-Protocol Analysis Set due to a large number of patients who discontinued the study (lack of assessments of iron exchange parameters at visits) and deviations from the Protocol affecting the assessment of efficacy parameters. Because of that, the additional efficacy analysis in the Per-Protocol Analysis Set was not performed.
Time Frame: Screening, Week (Wk) 4, Wk 8, Wk 12, Wk 16, Wk 20, Wk 24, Wk 28, Wk 32, Wk 36, Wk 40, Wk 44, Wk 48, Wk 52
Population: Full Analysis Set included all patients of the Safety Analysis Set with available baseline data & data obtained at follow-up visits &/or final visit, for evaluation of at least 1 efficacy parameter. Statistical analysis was not performed due to large number of patients discontinuing & thus lack of assessments of iron exchange parameters at visits.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Serum Ferritin Level ≥ 1,000 μg/l | Serum Ferritin Level < 1,000 μg/l
Number analyzed (Participants) | 10 | 5
ng/ml
  Screening | 2866.14 (1460.13) | 769.02 (230.36)
  Week 0 | 2895.62 (1245.81) | 727.68 (299.61)
  Week 4: number analyzed (Participants) | 9 | 4
  Week 4 | 2089.62 (638.29) | 640.75 (292.14)
  Week 8: number analyzed (Participants) | 9 | 5
  Week 8 | 2498.58 (1165.94) | 623.14 (223.27)
  Week 12: number analyzed (Participants) | 6 | 5
  Week 12 | 2262.12 (916.65) | 653.62 (311.72)
  Week 16: number analyzed (Participants) | 7 | 5
  Week 16 | 2164.01 (886.93) | 647.58 (225.28)
  Week 20: number analyzed (Participants) | 8 | 4
  Week 20 | 2054.23 (729.14) | 646.80 (147.73)
  Week 24: number analyzed (Participants) | 6 | 4
  Week 24 | 1710.67 (653.13) | 680.08 (182.24)
  Week 28: number analyzed (Participants) | 6 | 3
  Week 28 | 1446.07 (395.17) | 526.17 (122.40)
  Week 32: number analyzed (Participants) | 6 | 3
  Week 32 | 1626.28 (689.86) | 687.37 (114.47)
  Week 36: number analyzed (Participants) | 6 | 3
  Week 36 | 1709.07 (1153.94) | 699.13 (217.38)
  Week 40: number analyzed (Participants) | 6 | 3
  Week 40 | 1897.05 (1107.95) | 717.33 (306.63)
  Week 44: number analyzed (Participants) | 5 | 3
  Week 44 | 1301.80 (460.31) | 661.13 (267.15)
  Week 48: number analyzed (Participants) | 3 | 3
  Week 48 | 1740.00 (1493.24) | 709.50 (305.32)
  Week 52: number analyzed (Participants) | 1 | 3
  Week 52 | 1288.80 (NA) — N/A = not enough participants to calculate the standard deviation | 655.07 (277.98)

2. Primary Outcome: Change in Transferrin Saturation With Iron (TSI) Values
Description: Mean percentage change from baseline in transferrin saturation with iron was summarized descriptively for all on-treatment study visits.
Time Frame: Screening, Week (Wk) 4, Wk 8, Wk 12, Wk 16, Wk 20, Wk 24, Wk 28, Wk 32, Wk 36, Wk 40, Wk 44, Wk 48, Wk 52
Population: Full Analysis Set (FAS) included all patients of the Safety Analysis Set with the available baseline data, as well as data obtained at follow-up visits and/or the final visit, for evaluation of at least one efficacy parameter.
Measure: Mean (Standard Deviation); unit: Percentage of saturation
Arm/Group | Serum Ferritin Level ≥ 1,000 μg/l | Serum Ferritin Level < 1,000 μg/l
Number analyzed (Participants) | 10 | 5
Percentage of saturation
  Screening | 88.80 (10.01) | 53.70 (10.28)
  Week 0: number analyzed (Participants) | 9 | 4
  Week 0 | 87.19 (10.49) | 54.88 (14.50)
  Week 4: number analyzed (Participants) | 10 | 4
  Week 4 | 73.37 (8.55) | 50.10 (14.14)
  Week 8: number analyzed (Participants) | 9 | 5
  Week 8 | 72.68 (9.49) | 49.54 (17.12)
  Week 12: number analyzed (Participants) | 8 | 5
  Week 12 | 72.43 (5.98) | 49.04 (10.15)
  Week 16: number analyzed (Participants) | 7 | 4
  Week 16 | 68.60 (9.21) | 52.78 (9.21)
  Week 20: number analyzed (Participants) | 8 | 4
  Week 20 | 68.14 (19.64) | 50.65 (11.45)
  Week 24: number analyzed (Participants) | 6 | 4
  Week 24 | 74.30 (11.79) | 5.90 (5.59)
  Week 28: number analyzed (Participants) | 4 | 3
  Week 28 | 65.05 (7.57) | 52.67 (12.49)
  Week 32: number analyzed (Participants) | 6 | 3
  Week 32 | 75.75 (12.98) | 49.90 (11.96)
  Week 36: number analyzed (Participants) | 5 | 3
  Week 36 | 65.94 (13.87) | 47.83 (4.91)
  Week 40: number analyzed (Participants) | 6 | 3
  Week 40 | 66.05 (9.51) | 43.07 (2.57)
  Week 44: number analyzed (Participants) | 5 | 3
  Week 44 | 69.22 (16.95) | 33.27 (9.63)
  Week 48: number analyzed (Participants) | 3 | 3
  Week 48 | 71.07 (12.87) | 44.20 (1.39)
  Week 52: number analyzed (Participants) | 2 | 3
  Week 52 | 83.40 (11.74) | 43.57 (4.09)

3. Primary Outcome: Change in Serum Total Iron-binding Capacity (TIBC)
Description: Mean change from baseline in serum total iron-binding capacity was summarized descriptively for all on-treatment study visits.
Time Frame: Screening, Week (Wk) 4, Wk 8, Wk 12, Wk 16, Wk 20, Wk 24, Wk 28, Wk 32, Wk 36, Wk 40, Wk 44, Wk 48, Wk 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μmol/l
Arm/Group | Serum Ferritin Level ≥ 1,000 μg/l | Serum Ferritin Level < 1,000 μg/l
Number analyzed (Participants) | 10 | 5
μmol/l
  Screening | 4.51 (9.34) | 66.68 (14.95)
  Week 0: number analyzed (Participants) | 10 | 4
  Week 0 | 49.98 (10.17) | 49.10 (5.73)
  Week 4: number analyzed (Participants) | 10 | 4
  Week 4 | 78.70 (20.93) | 49.00 (4.95)
  Week 8: number analyzed (Participants) | 9 | 5
  Week 8 | 73.90 (10.97) | 47.44 (5.09)
  Week 12: number analyzed (Participants) | 8 | 5
  Week 12 | 83.56 (19.86) | 47.20 (4.68)
  Week 16: number analyzed (Participants) | 7 | 4
  Week 16 | 85.31 (23.12) | 49.53 (8.03)
  Week 20: number analyzed (Participants) | 8 | 4
  Week 20 | 74.34 (18.95) | 48.63 (4.46)
  Week 24: number analyzed (Participants) | 6 | 4
  Week 24 | 81.90 (27.17) | 46.53 (5.82)
  Week 28: number analyzed (Participants) | 5 | 3
  Week 28 | 101.90 (23.71) | 45.97 (4.14)
  Week 32: number analyzed (Participants) | 6 | 3
  Week 32 | 72.85 (25.92) | 48.23 (2.05)
  Week 36: number analyzed (Participants) | 5 | 3
  Week 36 | 76.56 (19.13) | 47.53 (2.60)
  Week 40: number analyzed (Participants) | 6 | 3
  Week 40 | 83.50 (19.74) | 46.30 (4.49)
  Week 44: number analyzed (Participants) | 5 | 3
  Week 44 | 71.56 (23.95) | 44.10 (4.22)
  Week 48: number analyzed (Participants) | 3 | 3
  Week 48 | 74.30 (11.61) | 45.70 (5.57)
  Week 52: number analyzed (Participants) | 2 | 3
  Week 52 | 67.10 (26.87) | 46.77 (5.39)

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 376 days.
Arm/Group | Serum Ferritin Level ≥ 1,000 μg/l | Serum Ferritin Level < 1,000 μg/l
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 4/10 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Serum Ferritin Level ≥ 1,000 μg/l (N=10) | Serum Ferritin Level < 1,000 μg/l (N=5)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Blood creatine increased (Investigations) | 2 (2) | 0 (0)
Weakness (General disorders) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety